CLINICAL TRIAL: NCT00211224
Title: Phase 3 Study of Riluzole in Multiple System Atrophy (MSA) and Progressive Supranuclear Palsy (PSP) (Parkinson's Plus Syndromes)
Brief Title: Neuroprotection and Natural History in Parkinson's Plus Syndromes (NNIPPS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); University of Ulm (Other); Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QLG1-2000-01262; European Commission; QLG1-2000-01262
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-09

CONDITIONS: Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: multiple system atrophy; progressive supranuclear palsy; riluzole; MSA; PSP
MeSH Terms: conditions — Multiple System Atrophy; Supranuclear Palsy, Progressive | interventions — Riluzole

INTERVENTIONS:
Drug: Riluzole

SUMMARY:
NNIPPS is a clinical trial of riluzole (a drug previously shown to slow down the rate of progression og amyotrophic lateral sclerosis-ALS; Lou Gehrig's disease) involving nearly 800 people diagnosed with the 'parkinson plus' syndromes of multiple system atrophy (MSA) and progressive supranuclear plasy (PSP). In addition to showing whether riluzole is helpful in MSA and PSP, NNIPPS will improve criteria for making an accurate and early diagnosis, for assessing the rate of progression, and will advance understanding of the biology of these disabling and progressive neurodegenerative diseases.

DETAILED DESCRIPTION:
Multiple System Atrophy (MSA) and Progressive Supranuclear Palsy (PSP) often present as akinetic-rigid syndromes and in the early stages are difficult to differentiate in the clinic. Current Consensus Diagnostic Criteria based on retrospective studies have high specificity but low sensitivity. The NNIPPS study is an EU-funded multinational (France, UK, Germany) multi-centre academic-led project with four main aims. The first aim is to test the hypothesis that riluzole, which may have generic neuroprotective properties, reduces the risk of death and improves function and quality of life (QL) in patients with MSA and PSP- 'parkinson's plus syndromes'. The second aim is to identify prognostic factors for survival and functional deterioration, and to develop and validate functional rating scales prospectively. The third aim is to investigate MRI, cognitive, pathological and genetic aspects of these disorders in relation to disease progression and pathogenesis. The fourth aim is to understand the impact of these diseases on the QL of patients and carers and to identify the health costs of treatment.

The study is designed as a randomised, stratified, controlled trial of the efficacy and safety of riluzole (up to 200mg daily) versus placebo in MSA and PSP. The primary outcome measure is survival at 36 months. Power calculations suggested that we would need to recruit ~400 patients into each stratum (MSA, PSP) in order to detect a reduction in the relative risk (RR) of death at 36 months with 80% power and two-sided a=0.05. Using modified consensus criteria (to provide greater sensitivity) we recruited 766 patients (363 PSP, 404 MSA) over 2 years (1999-2001). The first patients recruited are about to enter the open-label study. The final analysis of the primary efficacy measure is planned for December 2005. Secondary outcome measures include safety, rate of change in UPDRS and other rating scales including a parkinson's plus symtoms rating scale (PPSS), changes in cognitive function assessed using the Mattis Dementia Rating Scale, the Frontal Assessment Battery, The Bushke Selective Reminding Test, The Neuropsychiatric Inventory, and other tests of memory and executive function. QL and Health economic data is collected using the SF36 and a Client Service Receipt Inventory (CSRI). Assessments are made at 6 monthly intervals. Standardised MRI has been acquired in ~70% of cases at entry and will be repeated at 36 months where possible. DNA has been collected from ~75% of cases. 100 brains have been donated and are being analysed using a standardised protocol.

ELIGIBILITY:
Inclusion Criteria:

* akinetic rigid syndrome plus clinical criteria for MSA or PSP

Exclusion Criteria:

* Idiopathic Parkinson's disease
* Other neurological or serious medical disorders
* Unable to give informed consent
* dementia
* liver damage
* women of child bearing age unable to use effective method of contraception

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2000-04; Study Completion 2004-11

PRIMARY OUTCOMES:
survival

SECONDARY OUTCOMES:
functional measures (UPDRS, Parkinson's Plus Scale)
Change in MRI abnormalities
Cognitive changes

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Leigh, PhD FRCP, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, King's College London, London, London, United Kingdom

REFERENCES:
- [Derived] Payan CA, Viallet F, Landwehrmeyer BG, Bonnet AM, Borg M, Durif F, Lacomblez L, Bloch F, Verny M, Fermanian J, Agid Y, Ludolph AC, Leigh PN, Bensimon G; NNIPPS Study Group. Disease severity and progression in progressive supranuclear palsy and multiple system atrophy: validation of the NNIPPS--Parkinson Plus Scale. PLoS One. 2011;6(8):e22293. doi: 10.1371/journal.pone.0022293. Epub 2011 Aug 4. PMID 21829612
- [Derived] Rolland Y, Verin M, Payan CA, Duchesne S, Kraft E, Hauser TK, Jarosz J, Deasy N, Defevbre L, Delmaire C, Dormont D, Ludolph AC, Bensimon G, Leigh PN; NNIPPS Study Group. A new MRI rating scale for progressive supranuclear palsy and multiple system atrophy: validity and reliability. J Neurol Neurosurg Psychiatry. 2011 Sep;82(9):1025-32. doi: 10.1136/jnnp.2010.214890. Epub 2011 Mar 8. PMID 21386111
- [Derived] Al-Chalabi A, Durr A, Wood NW, Parkinson MH, Camuzat A, Hulot JS, Morrison KE, Renton A, Sussmuth SD, Landwehrmeyer BG, Ludolph A, Agid Y, Brice A, Leigh PN, Bensimon G; NNIPPS Genetic Study Group. Genetic variants of the alpha-synuclein gene SNCA are associated with multiple system atrophy. PLoS One. 2009 Sep 22;4(9):e7114. doi: 10.1371/journal.pone.0007114. PMID 19771175
- [Derived] Bensimon G, Ludolph A, Agid Y, Vidailhet M, Payan C, Leigh PN; NNIPPS Study Group. Riluzole treatment, survival and diagnostic criteria in Parkinson plus disorders: the NNIPPS study. Brain. 2009 Jan;132(Pt 1):156-71. doi: 10.1093/brain/awn291. Epub 2008 Nov 23. PMID 19029129